CLINICAL TRIAL: NCT02526979
Title: A Multicentre, Open-Label, Single Dose, Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Mirabegron Oral Suspension in Pediatric Subjects From 3 to Less Than 12 Years of Age With Neurogenic Detrusor Overactivity (NDO) or Overactive Bladder (OAB)
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Mirabegron Oral Suspension in Pediatric Subjects From 3 to Less Than 12 Years of Age With Neurogenic Detrusor Overactivity (NDO) or Overactive Bladder (OAB)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-203; 2015-000700-26 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder; Neurogenic Detrusor Overactivity
Keywords: OAB; overactive bladder; Myrbetric; neurogenic detrusor overactivity; Betanis; Myrbetriq; NDO; YM178; mirabegron; Betmiga
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mirabegron (Experimental): single dose
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: Myrbetriq; Myrbetric; Betanis; YM178; Betmiga

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK) of mirabegron oral suspension after single dose administration in children with neurogenic detrusor overactivity (NDO) or overactive bladder (OAB).

This study will also evaluate the safety and tolerability as well as the acceptability and palatability of mirabegron oral suspension after single dose administration in children with NDO or OAB.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female from 3 to less than 12 years of age.
* Subject has a documented diagnosis according to the International Children's Continence Society (ICCS) criteria of:

  * NDO, or
  * Idiopathic OAB
* Subject's weight/height:

  * Subject must have a body weight of ≥ 15.0 kg
  * For NDO: subject is not suffering from malnutrition or is not grossly overweight, in the opinion of the Investigator
  * For OAB: subject's weight and height are within the normal percentiles (3rd to 97th percentile) according to Centers for Disease Control and Prevention (CDC) growth charts.
* Subject is able to swallow the study medication in accordance with the protocol.
* Subject and subject's parent(s)/legal guardian agree that the subject will not participate in another interventional study while on treatment.
* Subject and subject's parent(s)/legal guardian are willing and able to comply with the study requirements and with the concomitant medication restrictions.
* Female subject must:

  * Be of non-childbearing potential: Clearly pre-menarchal or in the judgment of the Investigator is pre-menarchal.
  * Or the following inclusion criteria are to be followed, if applicable (rare cases): Female subject that reached puberty must: Agree not to try to become pregnant during the study and for 28 days after the final study drug administration, And have a negative urine pregnancy test predose Day 1, And, if heterosexually active agree to consistently use 2 forms of highly effective form of birth control starting at screening and throughout the study period and for28 days after the final study drug administration.

Exclusion Criteria:

* Subject has a known history of QTc prolongation or risk of QT prolongation (e.g. hypokalemia, family history of Long QT Syndrome) and/or QTcB of > 460 ms.
* Subject has a (mean) resting pulse rate > 99th percentile [Fleming et al, 2011].
* Subject has any clinically significant ECG (electrocardiogram) abnormality.
* Subject has established hypertension and a systolic or diastolic blood pressure greater than the 99th percentile of the normal range determined by sex, age and height, plus 5mmHg [NIH 2005].
* Subject has any clinically significant or unstable medical condition or disorder which, in the opinion of the Investigator, precludes the subject from participating in the study.
* Subject has current, untreated constipation (or fecal impaction for NDO subjects). If the constipation is being consistently treated for the last month, the subject can be included.
* Subject has been administered intradetrusor botulinum toxin injections; except if given > 4 months prior to screening and symptoms reappeared comparable to those before botulinum toxin injections.
* Subject has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than or equal to 2 times the ULN or total bilirubin greater than or equal to 1.5 times the ULN.
* Subject has severe renal impairment (estimated glomerular filtration rate < 30 mL/min (Larsson)).
* Subject has any other clinically significant out of range results of urinalysis, biochemistry or hematology.
* Subject has a history or current diagnosis of any malignancy.
* Subject has known or suspected hypersensitivity to mirabegron, other ß3-agonists, any of the excipients used in the mirabegron oral suspension formulation or previous severe hypersensitivity to any drug.
* Subject meets any of the contra indications or precautions for use of mirabegron listed in the Investigator's Brochure (IB).
* Subject has used mirabegron within 12 days of the planned Reference Day (Day -4 to Day -1).
* Subject requires ongoing treatment with any of the following prohibited medications:

  * Any anticholinergic/antimuscarinic drugs within 5 half-lives prior to planned Reference Day (Day -4 to Day -1).
  * Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index (such as thioridazine, flecainide, propafenone, imipramine, desipramine) and sensitive P-gp substrates (such as digoxin, dabigatran) within 5 half-lives prior to the planned Reference Day (Day -4 to Day -1).
  * Any moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers including natural and herbal remedies (such as itraconazole, rifampicin, phenytoin, carbamazepine, St. John's Wort, grapefruit, Seville orange) within 4 weeks (inducers only) or 5 half-lives (inhibitors only) prior to the planned Reference Day (Day -4 to Day -1).
* Subject has participated in another clinical trial and/or has taken an investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to the planned Reference Day (Day -4 to Day -1).
* Subject's parent(s)/legal guardian is an employee of the Astellas Group, any Contract Research Organization (CRO) involved, or the Investigator site executing the study.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of mirabegron in plasma: Cmax | Days 1 - 7
  Maximum concentration (Cmax)
Pharmacokinetics of mirabegron in plasma: AUCinf | Days 1 - 7
  Area under the curve from time zero to infinity (AUCinf)
Pharmacokinetics of mirabegron in plasma: tmax | Days 1 - 7
  The time after dosing when Cmax occurs (tmax)
Pharmacokinetics of mirabegron in plasma: t1/2 | Days 1 - 7
  Apparent Terminal Elimination Half-life (t1/2)

SECONDARY OUTCOMES:
Safety profile as assessed by adverse events, clinical laboratory evaluations, vital signs and electrocardiograms (ECG) | Up to Day 7
  Clinical laboratory evaluations include hematology, biochemistry and urinalysis.
Safety as assessed by post-void residual volume (PVR) | Day 1
Acceptability and Palatability as assessed by taste and acceptance of the suspension (5-point scale) | Day 1
  5-point scale consists of 3 questions ranging in score from 0=Really Bad to 4=Really Good.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (3):
- Denmark (2):
  - Site DK45002, Aalborg
  - Site DK45001, Aarhus
- Site PL48001, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;178-CL-203